CLINICAL TRIAL: NCT04306965
Title: Apremilast 30 mg BID Combined With Dupilumab for the Treatment of Recalcitrant Moderate-to-Severe Atopic Dermatitis
Brief Title: Apremilast 30 mg Twice Daily (BID) Combined With Dupilumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13305
Record Dates: First submitted 2020-03-04; First posted 2020-03-13 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apremilast (Experimental): Apremilast will be administered to patients as 30 mg oral tablets taken twice daily for 24 weeks. An initial 5-day titration will be implemented to improve tolerability.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 30 mg twice daily (BID)
  Other Names: Otezla

SUMMARY:
Open label phase 2 investigational study of efficacy and safety of apremilast 30 mg twice a day (BID) in chronic atopic dermatitis when added to the FDA approved treatment dupilumab for atopic dermatitis that is not providing adequate clinical responses.

DETAILED DESCRIPTION:
The purpose of this study is to determine if apremilast as a combined treatment for atopic dermatitis will provide increased efficacy outcomes in subjects who are currently using the FDA approved therapy of dupilumab but have responded only partially or inadequately to this therapy. Our hypothesis is that adding apremilast will allow patients to go from an inadequate response to dupilumab to an adequate response defined as an Investigator Global Assessment (IGA) of 0 (clear) or 1 (almost clear).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent indicating the subject has been informed of all aspects of the study
2. Subject is willing and able to comply with treatment plan, study drug administration, and study protocol requirements
3. Subject has a documented clinical diagnosis of chronic atopic dermatitis for at least 6 months prior to screening visit and is a candidate for systemic therapy
4. Subjects must fulfill criteria outlined in the following clinical categories:

   * Subjects must be currently using and experiencing an inadequate response to dupilumab which is FDA approved for the treatment of moderate to severe atopic dermatitis. An inadequate response is defined as an IGA of 2 or more.
   * At the time of screening, subject must have a partial or inadequate response to their current treatment regimen. A partial or inadequate response at screening is defined as having both of the following:
   * Not having achieved an Investigator's Global Assessment score of 0 (clear) or 1 (almost clear).
   * Subjects must be on dupilumab for at least 12 weeks and willing to continue on dupilumab on a stable dose (40 mg weekly or every other week) while also receiving the study drug
5. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options
6. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on study medication and for at least 28 days after the last dose of study medication
7. If receiving concomitant medications for any reason, must be on a stable regimen and willing to stay on a stable regimen. This includes emollients, which should stay stable throughout the study

Exclusion Criteria:

1. Prior hypersensitivity reaction or exposure to apremilast 2. Untreated or unstable depression or suicidality, including prior history of suicide attempt at any time in the subject's lifetime prior to Baseline Visit or major psychiatric illness requiring hospitalization within 3 years prior to Baseline Visit. Depression and suicidality will be assessed through standard-of-care questioning 3. Other than atopic dermatitis, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled 4. Any condition, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study 6. Pregnant or lactating females 7. Concomitant therapy with CYP450 enzyme inducers (e.g., rifampin, phenobarbital, carbamazepine, phenytoin), which may cause loss of efficacy of apremilast.

8. Prolonged sun exposure or use of tanning booths, which may confound the ability to interpret data from the study.

9. Active substance abuse or a history of substance abuse within 6 months prior to Screening. Subjects will be asked about any history of substance use using standard of care questioning.

10. Malignancy or history of malignancy, except for:

* treated [i.e., cured] basal cell or squamous cell in situ skin carcinomas;
* treated [i.e., cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.

  11. Use of dupilumab in combination with any other systemic immunosuppressant medication within 4 weeks prior to randomization or 5 pharmacokinetic/pharmacodynamic half lives, whichever is longer.

  12. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rosmarin, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast: Apremilast will be administered to patients as 30 mg oral tablets taken twice daily for 24 weeks. An initial 5-day titration will be implemented to improve tolerability.
  Apremilast: 30 mg BID
Period: Overall Study
Arm/Group | Apremilast
Started | 10
Completed | 4
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (21.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
weight in kg [Mean (Standard Deviation); unit: kilograms] | 86.38 (19.0)
concomitant topical steroid use [Count of Participants; unit: Participants] | 4
time on dupilumab therapy [Mean (Standard Deviation); unit: months] | 20.3 (14.3)
% patients with asthma [Count of Participants; unit: Participants] | 8
% patients with allergic rhinitis [Count of Participants; unit: Participants] | 8
% patients with food allergy [Count of Participants; unit: Participants] | 6
mean duration of atopic dermatitis [Mean (Standard Deviation); unit: years] | 18.6 (10.2)
prior atopic dermatitis treatments , % [Count of Participants; unit: Participants]
  topical corticosteroids | 10
  topical calcineurin inhibitor | 7
  immunosuppressants | 7
  phototherapy | 1
  prednisone | 6
  topical phosphodiesterase-4 inhibitor | 5
Investigator Global Assessment Score [Count of Participants; unit: Participants] — Investigator Global Assessment (IGA) Scale for Atopic Dermatitis consists of 5 severity scores ranging from 0 - 4. 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), 4 (severe).
  Participants
    IGA score 2 (Mild) | 3
    IGA score 3 (Moderate) | 7
baseline Body Surface Area (BSA), % [Mean (Standard Deviation); unit: % percentage of body surface area] | 9.99 (6.3)
Baseline Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: score on a scale] — 10-item questionnaire that measures how much the subjects' skin disease has affected their quality of life over the past week. Total score range 0 to 30, a score equal to zero (0) represents no impact and a score equal to thirty (30) represents severe impact on quality of life
  score on a scale | 7.6 (5.4)
Baseline Numerical Rating Scale (NRS) pruritus [Mean (Standard Deviation); unit: score on a scale] — zero (0) to ten (10) numerical rating scale, zero equals no itch and ten equals worst itch imaginable.
  score on a scale | 5.0 (2.4)
Baseline Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: score on a scale] — score ranges from zero (0) to seventy- two (72), 0 indicates no active eczema / atopic dermatitis, max score 72 indicates severe eczema involvement of all body regions
  score on a scale | 7.4 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve an Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16.
Description: Clinical improvement in a patient's eczematous lesions corresponds with a decrease in IGA, and a score of 0 (clear) or 1 (almost clear) is considered a significant clinical response.
Time Frame: week 16
Population: An intention-to-treat analysis was performed using last observation carried forward and included all enrolled patients who received apremilast at Week 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 10
Participants | 2

2. Secondary Outcome: Percentage of Subjects Achieving Body Surface Area Less Than 3% at Week 16
Time Frame: Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 10
Participants | 4

3. Secondary Outcome: Body Surface Area (BSA) Involvement
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Apremilast
Number analyzed (Participants) | 10
percentage of BSA | 5.5 (3.8)

4. Secondary Outcome: Body Surface Area (BSA) Involvement
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 10
percent change | -37.6 (26.6)

5. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: 10-item questionnaire that measures how much the subjects' skin disease has affected their quality of life over the past week. Total score range 0 to 30, a score equal to zero (0) represents no impact and a score equal to thirty (30) represents severe impact on quality of life.
Time Frame: baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 10
score on a scale | 3.7 (3.4)

6. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: as for outcome 5
Time Frame: baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 10
percent change | -36.9 (54.8)

7. Secondary Outcome: Numerical Rating Scale (NRS) Pruritus Scale
Description: zero (0) to ten (10) numerical rating scale, zero equals no itch and ten equals worst itch imaginable.
Time Frame: Baseline - Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 10
score on a scale | 2.9 (2.4)

8. Secondary Outcome: Numerical Rating Scale (NRS) Pruritus Scale
Description: zero (0) to ten (10) numerical rating scale, zero equals no itch and ten equals worst itch imaginable.
Time Frame: Baseline - Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 10
percent change | -45.9 (17.8)

9. Secondary Outcome: Eczema Area and Severity Index (EASI) Score
Description: score ranges from zero (0) to seventy- two (72), 0 indicates no active eczema / atopic dermatitis, max score 72 indicates severe eczema involvement of all body regions.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 10
score on a scale | 4.4 (2.5)

10. Secondary Outcome: Eczema Area and Severity Index (EASI) Score
Description: as for outcome 9
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Apremilast
Number analyzed (Participants) | 10
percent change | -32.6 (42.6)

11. Other Pre Specified Outcome: Safety Analysis
Description: Safety and tolerability will be evaluated by tabulations of adverse events
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Baseline - week 24
Arm/Group | Apremilast
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=10)
Gastrointestinal (GI) disturbances (Gastrointestinal disorders) | 5 (5) — (nausea, diarrhea, indigestion)
Headache (General disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Limitations of this study include the open-label design, small sample size, high drop-out rate and concomitant use of existing atopic dermatitis (AD) medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04306965/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04306965/SAP_003.pdf